CLINICAL TRIAL: NCT04447235
Title: Randomized, Doubled-blind Phase II Trial Evaluating the Use of Ivermectin Plus Losartan for Prophylaxis of Severe Events in Cancer Patients With Recent Diagnosis of COVID-19
Brief Title: Early Treatment With Ivermectin and LosarTAN for Cancer Patients With COVID-19 Infection
Acronym: TITAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility analysis has demonstrated no difference between arms
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP 1677/20
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cancer; COVID; Coronavirus Infection
Keywords: cancer; covid-19; losartan; ivermectin
MeSH Terms: conditions — Neoplasms; Coronavirus Infections; COVID-19 | interventions — Ivermectin; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: doubled-blind and placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: Placebo (Placebo Comparator): Patients will receive ivermectin-placebo single dose on the day of confirmed diagnosis of COVID-19, followed by losartan-placebo daily for 15 days.
  Interventions: Drug: Placebo
- ARM B: Ivermectin plus losartan (Experimental): Patients will receive a single dose of 12mg of ivermectin on the day of the confirmed diagnosis of COVID-19, followed by losartan 50mg orally once daily for 15 consecutive days
  Interventions: Drug: Ivermectin; Drug: Losartan

INTERVENTIONS:
Drug: Placebo — Use of the combination of ivermectin-placebo plus losartan-placebo as early treatment for COVID-19 in cancer patients
  Arms: ARM A: Placebo
Drug: Ivermectin — Use of the combination of ivermectin plus losartan as early treatment for COVID-19 in cancer patients
  Arms: ARM B: Ivermectin plus losartan
Drug: Losartan — Use of the combination of ivermectin plus losartan as early treatment for COVID-19 in cancer patients
  Arms: ARM B: Ivermectin plus losartan

SUMMARY:
Ivermectin plus losartan as prophilaxy to severe events in patients with cancer with recent diagnosis of COVID-19

DETAILED DESCRIPTION:
This is a randomized, doubled-blind and placebo-controlled phase II study that will evaluate the efficacy of the early use of ivermectin plus losartan in cancer patients who present with recent diagnosis of COVID-19.

The trial will enroll 176 patients with previous diagnosis of active cancer (88 in each arm) and the aim of the study is to assess the efficacy of these drugs combination to decrease the incidence of COVID-19 severe complications. Patients will receive single dose ivermectin of 12mg after the confirmed diagnosis of COVID-19, followed by 15 days of losartan.

We believe that the association of anti-viral activity of the ivermectin plus the extracellular blockade of the receptor used by the virus will decrease the overall viremia and subsequently improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Ability to understand and sign informed consent
* Biopsy-proven diagnosis of previous cancer (solid or hematologic disease)
* Participants must be diagnosed with active malignancy, defined as the presence of metastatic disease; or patient undergoing curative treatment during cancer treatment, regardless of the therapeutic modality.
* Confirmed diagnosis of COVID-19 by the presence of a positive PCR test or positive serological test and / or diagnosis presumed by the presence of flu-like symptoms associated to suggestive findings on CT scan.
* ECOG performance status 0 to 2
* Patients must have an assessment of adequate organ function within 28 days prior to enrollment, evidenced by:

  * Hemoglobin ≥ 9.0 g / dL
  * Leukometry> 2,000 / mm3
  * Absolute neutrophil count ≥ 1,500 / mm3
  * Platelet count ≥ 100,000 / mm3
  * Creatinine clearance ≥ 30 mL / min. Creatinine clearance (CrCl) should be calculated according to the Cockcroft-Gault formula.
  * Total bilirubin <3 x the upper limit of normal (ULN), except for patients with known Gilbert's syndrome.
  * Aspartate aminotransaminase (AST) <3.0 x LSN.
  * Alanine aminotransaminase (ALT) <3.0 x ULN.

Exclusion Criteria:

* Currently taking an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin receptor blocker (ARB).
* Patients who presents with severe conditions at the time of diagnosis requiring ICU admission.
* Prior reaction or intolerance to an ARB or ACE inhibitor.
* Blood pressure less than 110/70 mmHg at presentation
* Potassium greater than 5.0 mEq / L
* Pregnancy or breastfeeding
* Prior reaction to Ivermectin.
* Patient currently enrolled in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of severe complications due COVID-19 infection | 28 days
  Incidence of severe complications due COVID-19 infection defined as need for ICU admission, need for mechanical ventilation, or death

SECONDARY OUTCOMES:
Incidence of Severe Acute Respiratory Syndrome | 28 days
  Severe Acute Respiratory Syndrome defined as oxygen saturation less than 93%
Incidence of Severe Acute Respiratory Syndrome | 28 days
  Severe Acute Respiratory Syndrome defined as respiratory rate higher than 24 incursion per minute
Adverse events | 28 days
  Incidence of hepatic toxicity (elevation of ALT, AST above the upper limit of normal, measured by U/L)
Adverse events | 28 days
  Incidence of hepatic toxicity (elevation of bilirubin above the upper limit of normal, measured by mg/dL)
Adverse events | 28 days
  Incidence of renal toxicity (elevation of serum creatinine levels above the upper limit of normal, measured by mg/dL)
Adverse events | 28 days
  Incidence of symptomatic postural hypotension, diagnosed by clinical assessment of reduction of > 20 mmHG of arterial systolic pressure after measurement in prone position and orthostatic position.
Overall survival | 28 days
  Death of any cause since protocol enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Exman, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo; Maria del Pilar Diz, MD, PhD, Study Director — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
no plan to share individual participant data